CLINICAL TRIAL: NCT07261943
Title: The Effect of Sexual Counseling Based on the BETTER Model on Sexual Function and Quality of Sexual Life in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Serap Kırıcı, Lecturer, Karamanoğlu Mehmetbey University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Karamanoğlu Mehmetbey Universi
Record Dates: First submitted 2025-09-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Sexual Behavior; Climactericum; Sexuality Education
Keywords: BETTER model; sexuality; sexual education
MeSH Terms: conditions — Sexual Behavior; Sexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- experimental group (Experimental): The group that received sexual education based on the BETTER model
  Interventions: Other: The group that received sexual education based on the BETTER model

INTERVENTIONS:
Other: The group that received sexual education based on the BETTER model — The women in the experimental group will be trained in groups of 5-6, in a designated classroom in the Department of Obstetrics and Gynecology at the relevant hospital, in four sessions, each lasting 45-60 minutes, with a one-week break. The training will utilize warm-up exercises, PowerPoint presentations, question-and-answer sessions, and discussions. All women in the training group will be given the opportunity to ask questions and express themselves. Evaluation of the training will be conducted through Q&A and verbal feedback from the women, and further training will be provided on the requested topics based on their questions.No intervention will be made to the women in the control group after the pre-tests.
  Arms: experimental group

SUMMARY:
Sexual life, an integral part of overall health, remains one of the most neglected, undervalued, and problematic areas within today's healthcare system Various management strategies exist for managing sexual dysfunction, including behavioral, psychological, and pharmacological strategies, and researchers have used education and counseling interventions for this purpose. One such intervention is the BETTER model, which aims to collaborate with individuals experiencing sexual difficulties to address their problems. Discussing sexuality with individuals experiencing sexual difficulties and providing counseling services will significantly benefit healthcare professionals in promoting safe sexual practices, identifying existing or potential sexual problems, and addressing these issues

ELIGIBILITY:
Inclusion Criteria:

* Women who are married, sexually active, and have a regular sexual life
* Who are literate
* Who are postmenopausal (the time period between one year after menopause and old age within the WHO's definition of postmenopause)
* Who are more than one year postmenopause
* Who are not over 65 years of age, which is considered the age limit by the WHO -Who agree to participate in the study
* Who have entered menopause naturally-Who have scored ≤26.55 on the FSFI scale

Exclusion Criteria:

* Being on Hormone Replacement Therapy (HRT) and not having stopped at least six months before the study
* Having entered early menopause (before the age of 40)
* Having a chronic systemic disease and/or a psychiatric health problem
* Having a disability that makes communication difficult, such as hearing or language impairment
* Having received any sexual education before or during the study

Ages: 41 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 90 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Measuring the impact of sexual counseling based on the BETTER model | two months
  After sexual counseling based on the BETTER model, the Female Sexual Function Index (FSFI) scale were administered to women in the experimental and control groups via face-to-face interviews. The administration time for each scale varied between 15 and 20 minutes.
  Changes in the Female Sexual Function Index (FSFI) scale were measured two months after sexual counseling based on the BETTER model.
  Female Sexual Function Index (FSFI) It was developed by Rosen et al. as a multidimensional scale comprising 19 items to evaluate female sexual function. The scale includes six subheadings, desire, arousal, lubrication, orgasm, satisfaction, and pain. Each title was scored between 0 or 1 and six. The lowest and highest scores are 2 and 36, respectively. Higher scores indicated better sexual function. The cut-off value of the scale was 26.55. A total FSFI score of ≤26.55, it indicates sexual dysfunction

SECONDARY OUTCOMES:
Measuring the impact of sexual counseling based on the BETTER model | two months
  After sexual counseling based on the BETTER model, the Sexual Quality of Life-Female (SQoL-F) scale were administered to women in the experimental and control groups via face-to-face interviews. The administration time for each scale varied between 15 and 20 minutes.
  Changes in the Female Sexual Quality of Life (SQoL-F) scales were measured two months after sexual counseling based on the BETTER model.
  Sexual Quality of Life-Female (SQoL-F): Developed by Symonds et al., with Turkish validity and reliability conducted by Tuğut and Gölbaşı. It is a 6-point Likert-type scale with 18 items. Respondents consider their sexual life over the past four weeks. Scores range from 18 to 108. Higher scores indicate better sexual quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Karamanoglu Mehmetbey University, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No